CLINICAL TRIAL: NCT04044521
Title: Promoting the Implementation of Clinical Guidelines for Opioid Prescribing in Primary Care Using Systems Consultation
Brief Title: Promoting Clinical Guidelines for Opioid Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-1276; R01DA047279 (NIH); A532007 (Other: UW Madison); SMPH/FAMILY MED/RES GRANTS (Other: UW Madison); Protocol Version 8/31/2020 (Other: UW Madison)
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-05

CONDITIONS: Opioid Use
Keywords: implementation; primary care; organizational change; Centers for Disease Control opioid prescribing guidelines; clinical guidelines; systems consultation

STUDY DESIGN:
Intervention Model Description: The intervention will assess outcomes at the clinic and prescriber level. Prescribers are the population of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Academic detailing only (Experimental): Clinicians will attend an educational meeting and receive audit and feedback reports for 18 months.
  Interventions: Other: Systems consultation
- Academic detailing+practice facilitation (Experimental): Clinicians of this group will attend an educational meeting and receive a monthly audit and feedback report for 18 months.
  At month 3, clinics will be randomized to receive practice facilitation. Clinics will be asked to follow-up with the facilitators via phone or video chat monthly for months 4-9, then quarterly for months 10-18.
  Interventions: Other: Systems consultation
- Academic detailing+practice facilitation+physician peer consul (Experimental): Clinicians will receive academic detailing at month 0 and practice facilitation at month 3. At month 9, clinics will be randomized to receive physician peer consulting. Clinicians of the clinics will meet up to 4 times, quarterly, with the physician peer consultant.
  Interventions: Other: Systems consultation
- Academic detailing+physician peer consulting (Experimental): Clinicians of this group will attend an educational meeting and will receive a monthly audit and feedback report for 18 months.
  At month 9, clinicians of the clinics will meet up to 4 times, quarterly, with the physician peer consultant.
  Interventions: Other: Systems consultation

INTERVENTIONS:
Other: Systems consultation — Systems consultation consists of three implementation strategies: academic detailing (AD), practice facilitation (PF), and physician peer consulting (PPC). Clinics will receive a combination of these strategies for 21 months.
  AD: Clinicians will attend an educational meeting that will detail the study and Center for Disease Control guidelines for opioid prescribing in primary care. Clinicians will then will get a monthly audit & feedback report on their prescribing.
  PF: clinics will be randomized to receive practice facilitation. Facilitators will meet with each clinic. Facilitators walk through the clinic, identify areas of opioid prescribing workflow improvement, conduct a nominal group technique with the change team, and set a Plan-Do-Study-Act cycle. Clinics will follow-up with the facilitators monthly.
  PPC: Clinicians of the clinics will meet quarterly with the physician peer consultant to discuss tough patient cases and panels regarding opioid prescribing.

SUMMARY:
This study aims to understand the optimal sequencing and combination of implementation strategies that specific types of clinics and prescribers need to adopt clinical guidelines for opioid prescribing. The pragmatic goal is to give health systems a tool they can use to predict which clinics and prescribers will benefit most from which sequence and combination of implementation strategies.

DETAILED DESCRIPTION:
The proposed study evaluates a sequence and combination of implementation strategies that is tailored to the needs of stakeholders at different levels (health system, clinic, and prescriber). We will deliver an adaptive version of systems consultation that progressively and adaptively drills down to offer more and more personalized levels of implementation support. The intervention starts with academic detailing, a systems-level strategy consisting of an expert-led training session plus distance-based follow up support. This strategy continues for the 21-month intervention for all clinics, but at 3 months, half of the clinics will be randomized to receive practice facilitation. Practice facilitation is a clinic-level strategy in which a highly-skilled external change agent helps clinics improve processes related to opioid prescribing. At 6 months, half of prescribers will be randomized to receive physician peer coaching. Physician peer coaching is a clinic-level strategy in which a physician expert gives one-on-one support to prescribers in managing their patients on long-term opioid therapy. These 3 discrete strategies will be delivered in a sequential, multiple-assignment randomized trial to 38 clinics from 2 Wisconsin health systems. The study has 3 specific aims:

1. Compare the effect over 21 months of (1). An adaptive systems consultation implementation strategy (intervention group) vs. (2). Academic detailing alone (control group) on average morphine milligram equivalent dose (the primary outcome).
2. Develop an assessment of contextual factors that influence the effectiveness of different implementation strategies. This aim will test 4 moderators and assess other factors that affect implementation. The goal is to develop a tool that decision-makers can use to predict which implementation strategies will be most effective in different settings.
3. Estimate the costs of delivering 4 different sequences and combinations of strategies, including the incremental cost effectiveness of adding facilitation and physician peer coaching. Results will help decision-makers weigh the costs and effects of using different implementation strategies.

ELIGIBILITY:
Inclusion Criteria:

Clinics will be eligible for the study if they:

* are a primary care clinic (non-pediatric primary care, internal medicine, or family medicine);
* have not received the systems consultation intervention;
* do not explicitly prohibit initiating opioid therapy;
* do not exceed the performance on key measures of guideline concordance (fewer than 80% of long-term opioid patients have treatment agreements and a urine drug screen in the past 12 months)

Prescribers will be eligible if they:

* are a primary care provider at the clinic;
* are not temporary providers who do not manage stable panels or patients;

While patients are not subjects of study, de-identified prescriber panel data will be used to assess outcome measures. To be included in the de-identified prescriber panel data, patients must:

* have a primary care provider at the clinic;
* are prescribed opioid therapy for at least 3 consecutive months;
* do not have a cancer diagnosis or are receiving hospice care.

Exclusion Criteria:

Clinics will be excluded if they are not a primary care clinic, have received the systems consultation intervention, prohibit initiating opioid therapy, or exceed the threshold on key measures of guideline concordance.

Prescribers will be excluded if they don't have prescribing privileges or are temporary providers who do not manage stable panels or patients.

De-identified prescriber panel data will be excluded from outcome measures if they do not have a primary care provider at the clinic, are not prescribed opioid therapy for at least 3 consecutive months, or have a cancer diagnosis or are receiving hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Quanbeck, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Bellin Health Systems, Green Bay, Wisconsin
  - UW Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification will be available to researchers for independent verification of study outcomes or to conduct subsequent clinical research, whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 9 months after publication of primary outcomes, and ending 3 years following publication.
Access Criteria: Proposals should be directed to PI Andrew Quanbeck at arquanbe@wisc.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- [Background] Quanbeck A, Almirall D, Jacobson N, Brown RT, Landeck JK, Madden L, Cohen A, Deyo BMF, Robinson J, Johnson RA, Schumacher N. The Balanced Opioid Initiative: protocol for a clustered, sequential, multiple-assignment randomized trial to construct an adaptive implementation strategy to improve guideline-concordant opioid prescribing in primary care. Implement Sci. 2020 Apr 25;15(1):26. doi: 10.1186/s13012-020-00990-4. PMID 32334632
- [Derived] Quanbeck A, Robinson J, Jacobson N, Li X, Hennessy-Garza R, Landeck J, Cohen A, Madden L, Pulvermacher A, Brown R. Strategies to Deimplement Opioid Prescribing in Primary Care: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2438325. doi: 10.1001/jamanetworkopen.2024.38325. PMID 39388183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study team focused outreach efforts toward clinics to build awareness about this study. An email was sent to clinic medical directors of the health system to instruct them how to opt-out if they wish to decline participation in the study and future contact from the study team. The study team enrolled 'providers' as participants and focused on clinic-level data.
Units Other Than Participants: Clinics
Groups:
- Academic Detailing Only: Clinicians will attend an educational meeting and receive audit and feedback reports for 18 months.
  Systems consultation: Systems consultation consists of three implementation strategies: academic detailing (AD), practice facilitation (PF), and physician peer consulting (PPC). Clinics will receive a combination of these strategies for 18 months.
  AD: Clinicians will attend an educational meeting that will detail the study and Center for Disease Control guidelines for opioid prescribing in primary care. Clinicians will then will get a monthly audit & feedback report on their prescribing.
  PF: clinics will be randomized to receive practice facilitation. Facilitators will travel to each clinics. Facilitators walk through the clinic, identify areas of opioid prescribing workflow improvement, conduct a nominal group technique with the change team, and set a Plan-Do-Study-Act cycle. Clinics will follow-up with the facilitators monthly.
  PPC: Clinicians of the clinics will meet quarterly with the physician peer consultant to discuss tough patient cases and panels regarding opioid prescribing.
- Academic Detailing+Practice Facilitation: Clinicians of this group will attend an educational meeting and receive a monthly audit and feedback report for 18 months.
  At month 3, clinics will be randomized to receive practice facilitation. Clinics will be asked to follow-up with the facilitators via phone or video chat monthly for months 4-6, then quarterly for months 7-18.
  Systems consultation: Systems consultation consists of three implementation strategies: academic detailing (AD), practice facilitation (PF), and physician peer consulting (PPC). Clinics will receive a combination of these strategies for 18 months.
  AD: Clinicians will attend an educational meeting that will detail the study and Center for Disease Control guidelines for opioid prescribing in primary care. Clinicians will then will get a monthly audit & feedback report on their prescribing.
  PF: clinics will be randomized to receive practice facilitation. Facilitators will travel to each clinics. Facilitators walk through the clinic, identify areas of opioid prescribing workflow improvement, conduct a nominal group technique with the change team, and set a Plan-Do-Study-Act cycle. Clinics will follow-up with the facilitators monthly.
  PPC: Clinicians of the clinics will meet quarterly with the physician peer consultant to discuss tough patient cases and panels regarding opioid prescribing.
- Academic Detailing+Practice Facilitation+Physician Peer Consul: Clinicians will receive academic detailing at month 0 and practice facilitation at month 3. At month 6, clinics will be randomized to receive physician peer consulting. Clinicians of the clinics will meet up to 4 times, quarterly, with the physician peer consultant.
  Systems consultation: Systems consultation consists of three implementation strategies: academic detailing (AD), practice facilitation (PF), and physician peer consulting (PPC). Clinics will receive a combination of these strategies for 18 months.
  AD: Clinicians will attend an educational meeting that will detail the study and Center for Disease Control guidelines for opioid prescribing in primary care. Clinicians will then will get a monthly audit & feedback report on their prescribing.
  PF: clinics will be randomized to receive practice facilitation. Facilitators will travel to each clinics. Facilitators walk through the clinic, identify areas of opioid prescribing workflow improvement, conduct a nominal group technique with the change team, and set a Plan-Do-Study-Act cycle. Clinics will follow-up with the facilitators monthly.
  PPC: Clinicians of the clinics will meet quarterly with the physician peer consultant to discuss tough patient cases and panels regarding opioid prescribing.
- Academic Detailing+Physician Peer Consulting: Clinicians of this group will attend an educational meeting and will receive a monthly audit and feedback report for 18 months.
  At month 6, clinicians of the clinics will meet up to 4 times, quarterly, with the physician peer consultant.
  Systems consultation: Systems consultation consists of three implementation strategies: academic detailing (AD), practice facilitation (PF), and physician peer consulting (PPC). Clinics will receive a combination of these strategies for 18 months.
  AD: Clinicians will attend an educational meeting that will detail the study and Center for Disease Control guidelines for opioid prescribing in primary care. Clinicians will then will get a monthly audit & feedback report on their prescribing.
  PF: clinics will be randomized to receive practice facilitation. Facilitators will travel to each clinics. Facilitators walk through the clinic, identify areas of opioid prescribing workflow improvement, conduct a nominal group technique with the change team, and set a Plan-Do-Study-Act cycle. Clinics will follow-up with the facilitators monthly.
  PPC: Clinicians of the clinics will meet quarterly with the physician peer consultant to discuss tough patient cases and panels regarding opioid prescribing.
Period: Overall Study
Arm/Group | Academic Detailing Only | Academic Detailing+Practice Facilitation | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Started | 60; 8 Clinics | 65; 8 Clinics | 66; 8 Clinics | 77; 8 Clinics
Completed | 60; 8 Clinics | 65; 8 Clinics | 66; 8 Clinics | 77; 8 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on clinic-level data, participant-level data not collected.
Units Other Than Participants: Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Academic Detailing Only | Academic Detailing+Practice Facilitation | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting | Total
Number analyzed (Participants) | 60 | 65 | 66 | 77 | 268
Number analyzed (Clinics) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — unknown and not applicable Population: Participant level data not collected
  years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — unknown and not applicable Population: unknown and not applicable
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
    Female | 0 | 0 | 0 | 0 | 0
    Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
    (all) |  |  |  |  | 0
Average MME per day for most recent 3 months [Mean (Standard Deviation); unit: morphine milligram equivalents per day] — morphine milligram equivalents (MME)
  morphine milligram equivalents per day | 44.9938 (22.4591) | 39.6526 (17.2418) | 36.6330 (15.7656) | 48.9800 (20.1475) | 43.3 (19.7)
Percent of patients with average MME greater than or equal to 90 mg/day [Mean (Standard Deviation); unit: percent of patients] | 0.1142 (0.1175) | 0.1033 (0.1014) | 0.0741 (0.0954) | 0.1326 (0.1080) | 0.109 (0.109)
Percent of patients with co-prescribed Benzodiazepine in the last quarter [Mean (Standard Deviation); unit: percent of patients] | 0.1600 (0.0920) | 0.1123 (0.0817) | 0.1351 (0.1097) | 0.1178 (0.1095) | 0.132 (0.1)
Percent of patients with urine drug screen in last 12 months [Mean (Standard Deviation); unit: percent of patients] | 0.3302 (0.2577) | 0.2555 (0.2343) | 0.2628 (0.2089) | 0.3276 (0.2087) | 0.298 (0.234)
Percent of patients with treatment in last 12 months [Mean (Standard Deviation); unit: percent of patients] | 0.3302 (0.1946) | 0.1316 (0.2047) | 0.1982 (0.1593) | 0.1341 (0.1711) | 0.16 (0.188)
Percent of patients with PHQ-8/9 depression screen in last 12 months [Mean (Standard Deviation); unit: percent of patients] | 0.2791 (0.1936) | 0.2464 (0.1584) | 0.2673 (0.2101) | 0.2346 (0.1563) | 0.258 (0.18)
Percent of patients with PEG-3 pain screen in last 12 months [Mean (Standard Deviation); unit: percent of patients] | 0.1234 (0.2070) | 0.0291 (0.0596) | 0.0073 (0.0157) | 0.0919 (0.1602) | 0.069 (0.151)

OUTCOME MEASURES:

1. Primary Outcome: Average Morphine Milligram Equivalent (MME) Per Day of Chronic Opioid Prescriptions of Clinics
Description: The average morphine milligram equivalent will be reported at the clinic level. Patients included in this outcome are those who are prescribed at least 3 opioid orders in the last 3 consecutive months.
  For a comparison of opioids doses, a conversion factors were developed to equate the many different opioids into one standard value. This standard value is based on morphine and its potency, referred to as morphine milligram equivalents (MME) or morphine equivalent doses (MED).
Time Frame: up to 30 months
Population: Outcome measure provides clinic-level data. Participants enrolled are providers.
Measure: Mean (Standard Deviation); unit: average MME/day
Units Other Than Participants: Clinics
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
Number analyzed (Clinics) | 8 | 8 | 8 | 8
average MME/day | 320.69 (11.80) | 372.33 (20.04) | 275.55 (16.78) | 455.62 (19.59)

2. Primary Outcome: Average Morphine Milligram Equivalent of Chronic Opioid Prescriptions of Prescribers
Description: The average morphine milligram equivalent will be reported at the prescriber level. Patients included in this outcome are those who are prescribed at least 3 opioid orders in the last 3 consecutive months.
Time Frame: up to 30 months
Population: Outcome measure provides prescriber-level data. Participants enrolled are providers.
Measure: Mean (Standard Deviation); unit: average MME/day
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
average MME/day | 39.65 (17.24) | 45.00 (22.46) | 36.63 (15.77) | 48.98 (20.15)

3. Secondary Outcome: Number of Eligible Clinics That Participated
Description: The number of eligible clinics that participated in the study.
Time Frame: up to 30 months
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
Number analyzed (Clinics) | 8 | 7 | 8 | 8
Clinics | 8 | 7 | 8 | 8

4. Secondary Outcome: Number of Clinicians Who Participated in the Study
Description: The number of eligible clinicians who participated in the study
Time Frame: up to 30 months
Measure: Number; unit: participants
Units Other Than Participants: clinics
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
Number analyzed (clinics) | 8 | 7 | 8 | 8
participants | 65 | 60 | 66 | 77

5. Secondary Outcome: Number of Patients at Clinics
Description: The total number of patients seen at clinics will be used to assess clinic size.
Time Frame: up to 30 months
Measure: Number; unit: patients
Units Other Than Participants: clinics
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
Number analyzed (clinics) | 8 | 7 | 8 | 8
patients | 2486 | 2427 | 2044 | 2021

6. Secondary Outcome: Number of Clinicians Who Attended the Intervention Meetings
Description: The number of clinicians who attended the meeting for practice facilitation, physician peer consulting, and follow-up meetings.
Time Frame: up to 30 months
Measure: Mean (Standard Deviation); unit: average participants
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
average participants | 6.118461538 (11.36059744) | 6.741935484 (18.26451613) | 6.228070175 (22.34556254) | 6.15 (28.32195122)

7. Secondary Outcome: Average Hours of Intervention Received Per Clinic
Description: The average time (in hours) of intervention that clinics received.
Time Frame: up to 30 months
Measure: Mean (Standard Deviation); unit: hours
Units Other Than Participants: Clinics
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
Number analyzed (Clinics) | 8 | 7 | 8 | 8
hours | 12.5 (17.5) | 4.571428571 (1.673469388) | 14.875 (31.609375) | 6.125 (9.609375)

8. Secondary Outcome: Average Hours of Intervention Received Per Prescriber
Description: The average time (in hours) of intervention that prescribers received. The average time the prescriber received the intervention (in hours) is the same amount of time as the average intervention time that each clinic receives, because our intervention is at the clinic level.
Time Frame: up to 30 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
hours | 12.5 (17.5) | 4.571428571 (1.673469388) | 14.875 (31.609375) | 6.125 (9.609375)

9. Secondary Outcome: Estimated Cost of Each Study Arm in US Dollars
Description: The estimated cost of each implementation sequence and combination in US dollars. The result is derived from the number of intervention hours calculated for each arm, multiplied by the average salary of the staff who gave the intervention (e.g., the facilitators, providers, and IT coordinator), referenced from publicly reported data (Medscape Family Medicine Physician Compensation Report).
Time Frame: up to 30 months
Measure: Number; unit: dollars
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
dollars | 7933.2 | 2307.84 | 9015 | 4399.32

10. Other Pre Specified Outcome: Quality Improvement Experience of the Clinics
Description: A assessment tool is under development to capture the quality improvement experience level of clinics.
Time Frame: up to 30 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Components of System-level Opioid Prescribing Policy of the Health Systems
Description: A list and count of the components of the participating health systems' opioid prescribing policy.
Time Frame: up to 30 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Adaptations Made to the Intervention During Intervention Period
Description: A list and count of adaptations that were made to the intervention during the intervention period will be documented.
Time Frame: up to 30 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Number of Patients of a Prescriber Who Have Chronic Opioid Prescriptions
Description: The number of patients who are prescribed at least 3 opioid orders in 3 consecutive months. The number will be reported at the prescriber level.
Time Frame: up to 30 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Number of Patients Completing Urine Drug Screens in the Past 12 Months
Description: Number of patients who are prescribed at least 3 opioid orders in 3 consecutive months, who have had a urine drug screen documented within the past 12 months.
Time Frame: up to 30 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Number of Patients Completing Screening for Mental Health and Substance Abuse Within the Past 12 Months
Description: Number of patients who are prescribed at least 3 opioid orders in 3 consecutive months, who have a Patient Health Questionnaire (PHQ-9) documented within the past 12 months. The study team is not administering the screening tool, data will be provided by Wisconsin Collaborative for Healthcare Quality (WCHQ).
  The PHQ-9 is a 9-question instrument given to patients in a primary care setting to screen for the presence and severity of depression. It is the 9-question depression scale from the Patient Health Questionnaire. Total score can range from 1-27. Interpretation of total scores is as follows:
  1-4=Minimal depression, 5-9=Mild depression, 10-14= Moderate depression, 15-19=Moderately severe depression, 20-27= Severe depression.
Time Frame: up to 30 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Number of Patients With Treatment Agreements Within the Past 12 Months
Description: The number of patients who are prescribed at least 3 opioid orders in 3 consecutive months, who have documented treatment agreements within the past 12 months.
Time Frame: up to 30 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Number of Patients With a Daily Morphine Milligram Equivalent Above 90 Milligrams
Description: The number of patients who are prescribed at least 3 opioid orders in 3 consecutive months and have a daily morphine milligram equivalent over 90 milligrams.
Time Frame: up to 30 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Number of Patients Who Are Co-prescribed Opioids and Benzodiazepines
Description: Number of patients who are prescribed at least 3 opioid orders in 3 consecutive months, who also have a concurrent benzodiazepine prescription.
Time Frame: up to 30 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Number of Emergency Room Visits and Hospitalizations Per Patient
Description: The number of hospital or emergency room visits per patient among patients who are prescribed at least 3 opioid orders in 3 consecutive months.
Time Frame: up to 30 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Number of Patients Who Attend Their Scheduled Clinic Visits
Description: The number of patients who are prescribed at least 3 opioid orders in 3 consecutive months, who attend their scheduled clinic visits.
Time Frame: up to 30 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Total Number of Patients in a Clinic Who Have Chronic Opioid Prescriptions
Description: The total number of patients who are prescribed at least 3 opioid orders in 3 consecutive months. The number will be reported at the clinic level.
Time Frame: up to 30 months
Population: In this outcome measure, we report the number of patients who are prescribed at least 3 opioid orders in 3 consecutive months at the clinic level.
Measure: Number; unit: patients
Units Other Than Participants: Clinics
Arm/Group | Academic Detailing+Practice Facilitation | Academic Detailing Only | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
Number analyzed (Participants) | 65 | 60 | 66 | 77
Number analyzed (Clinics) | 8 | 8 | 8 | 8
patients | 985 | 1175 | 681 | 925

22. Other Pre Specified Outcome: Average Morphine Milligram Equivalent of Patients Who Are Co-prescribed Opioids and Benzodiazepines
Description: The average morphine milligram equivalent of patients who are prescribed at least 3 opioid orders in 3 consecutive months at the clinic level.
Time Frame: up to 30 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: not applicable - clinic level data collected
Arm/Group | Academic Detailing Only | Academic Detailing+Practice Facilitation | Academic Detailing+Practice Facilitation+Physician Peer Consul | Academic Detailing+Physician Peer Consulting
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
All eligible clinics in two health systems were invited to participate. Clinics that volunteered may have been more motivated to change. Also, the interventions began in Feb. 2020 shortly before COVID forcing the implementation interactions to be done virtually rather than in person. In addition, the 2016 CDC guidelines that formed the basis of the intervention were the subject of considerable debate in the medical community and were revised in Feb. 2022, near the end of the intervention period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT04044521/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04044521/ICF_001.pdf